CLINICAL TRIAL: NCT01223911
Title: A Randomised, Double-blind, Placebo-controlled, Multiple Dose Trial of NNC 0151-0000-0000 in Subjects With Rheumatoid Arthritis
Brief Title: A Multiple Dose Trial of NNC 0151-0000-0000 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8209-3607; U1111-1116-2430 (Other: WHO); 2009-011791-30 (EudraCT Number)
Record Dates: First submitted 2010-10-14; First posted 2010-10-19 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: NNC 0151-0000-0000
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC 0151-0000-0000 — Multiple doses will be administered subcutaneously (under the skin), one dose once weekly during a three week period
  Arms: A
Drug: placebo — Multiple doses will be administered subcutaneously (under the skin), one dose once weekly during a three week period
  Arms: B

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety, tolerability and pharmacokinetics (at which rate the drug is eliminated from the body) of NNC 151-0000-0000 in subjects with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* CZ: Age between 18 and 65 years (both inclusive)
* A diagnosis of rheumatoid arthritis of at least three months before entry in trial
* Active rheumatoid arthritis (RA)
* Subjects are on stable doses of methotrexate (up to and including 25 mg/week) for at least 4 weeks before trial drug administration

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Body mass index (BMI) less than 18.0 or more than 38.0 kg/m2 (inclusive)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | at all scheduled visits (week 1 - week 11)

SECONDARY OUTCOMES:
Serum concentrations of NNC 151-0000-0000 | at 48 hours after all dose administrations

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (15):
- Novo Nordisk Investigational Site, Prague, Czechia
- Denmark (2):
  - Novo Nordisk Investigational Site, Frederiksberg
  - Novo Nordisk Investigational Site, Silkeborg
- Novo Nordisk Investigational Site, Budapest, Hungary
- Poland (4):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Elblag
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Poznan
- Romania (4):
  - Novo Nordisk Investigational Site, Bacau, Bacău
  - Novo Nordisk Investigational Site, Cluj-Napoca, Cluj
  - Novo Nordisk Investigational Site, Sfântu Gheorghe, Covasna
  - Novo Nordisk Investigational Site, Bucharest
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Burslem
  - Novo Nordisk Investigational Site, Newcastle upon Tyne
  - Novo Nordisk Investigational Site, Swansea

REFERENCES:
- [Result] Daniluk S, Skrumsager BK, Leszczynski P. Safety and tolerability of the anti-C5aR humanised monoclonal antibody NNC0151-0000 in patients with rheumatoid arthritis: A phase 2, randomised, double-blind, placebocontrolled, multiple-dose trial. EULAR (European League Against Rheumatism) 2014; Country: France City: Paris
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com